CLINICAL TRIAL: NCT03779867
Title: Acute Effects of Exercise on Breast Cancer Biomarkers (ACE) Study
Brief Title: Acute Exercise Intervention in Breast Cancer Survivors
Acronym: ACE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed per SRC low accrual policy.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RG1003977; NCI-2018-02831 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 8766 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — RE1-silencing transcription factor

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: All study personnel other than the statisticians and exercise physiologist will be masked to participant study arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (acute exercise) (Experimental): Participants undergo a moderate-intensity acute exercise bout over 45 minutes.
  Interventions: Behavioral: Exercise Intervention; Other: Biomarker Analysis; Other: Questionnaire Administration
- Arm II (rest) (Active Comparator): Participants rest by sitting for 45 minutes.
  Interventions: Other: Resting; Other: Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Exercise Intervention — Undergo acute exercise
  Arms: Arm I (acute exercise)
Other: Resting — Seated resting
  Other Names: Rest
  Arms: Arm II (rest)
Other: Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how a 45-minute bout of acute exercise in women with a history of breast cancer can affect factors associated with breast cancer and help doctors learn more about how exercise can help prevent breast cancer.

In an earlier part of the study, investigators looked at the effects of the same intervention in women without a history of cancer.

DETAILED DESCRIPTION:
OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants undergo a moderate-intensity acute exercise bout over 45 minutes.

ARM II: Participants rest by sitting for 45 minutes.

EXTENSION: After completion of initial study recruitment and data collection, an extension was approved in 2023.

EXTENSION OUTLINE: Participants are randomized to 1 of 2 arms.

EXTENSION ARM I: Participants exercise on a stationary bike for 45 minutes.

EXTENSION ARM II: Participants rest by sitting for 45 minutes.

ELIGIBILITY:
Current Inclusion Criteria (for Extension participants):

* Female
* History of Stage 0-IIIc breast cancer, diagnosed within the last 5 years
* Completed primary treatment at least 6 months ago
* Able to attend 2 clinic visits at the Fred Hutch Prevention Center for approximately 2.5 hours at a time
* Aged 36-75 years. Younger women will be excluded because a sizable proportion may remain premenopausal and will resume menstruation within 2 years of chemotherapy completion.
* Postmenopausal (no menstrual periods in the previous 12 months either naturally, or as a consequence of treatment)
* All race and ethnic groups are eligible for the study
* Able to perform all study requirements, including attendance at clinic visits and capable of responding to questionnaires and clinic and exercise facility instructions in English
* Willing to consent to release of medical records for their breast cancer diagnosis and treatment
* If a patient has received a cardiotoxic therapy (e.g., Adriamycin, Herceptin), clearance of their oncologist to participated in this study will be required.

Completed Inclusion Criteria (for participants enrolled prior to Extension portion of study):

* Resident in greater Seattle metropolitan area (King County), Pierce or Snohomish Counties
* Healthy
* Able to perform all study requirements, including attendance at clinic visits and capable of responding to questionnaires and clinic and exercise facility instructions in English
* Willing to be randomized
* Capable of providing informed consent

Current Exclusion Criteria (for Extension participants):

* Family history of breast cancer
* If known, BRCA 1/2 mutation carrier
* If known, Li-Fraumeni Syndrome
* Personal history of cancer other than breast: exceptions are non-melanoma skin cancer and cervical neoplasia (CIN)
* Serious health conditions including diabetes, renal disease (e.g., chronic kidney disease), liver disease (e.g., cirrhosis, chronic liver failure), chronic lung disease (COPD, moderate or severe persistent asthma), auto-immune disease requiring oral or inhaled medication, congestive heart failure, or other condition likely to interfere with ability to exercise at moderate levels and undergo biosampling, or likely to interfere with study outcomes.
* Fasting glucose fingerstick >126 mg/dL
* Taking any medications to treat high blood sugar such as metformin
* Contraindications for exercise testing (29) including: recent (within 6 months) cardiac event (MI, pulmonary edema, myocarditis, pericarditis), unstable angina, uncontrolled arrhythmia, third degree heart block, left bundle branch block, acute congestive failure, recent (within 6 months) pulmonary/systemic embolus, severe electrolyte abnormality, deep vein thrombosis, uncontrolled hypertension (systolic > 200, diastolic > 100), orthostatic hypotension, moderate/severe aortic stenosis, uncontrolled arrhythmia, uncontrolled congestive heart failure, history of cardiac arrest or stroke, or as assessed by the physician assistant during the physical exam.
* History of clotting disorders
* Unable or unwilling to stop aspirin or NSAIDs for 48 hours before and after the procedure
* Allergy to anesthetics or local anesthetics
* Long term use of warfarin or similar medications
* Use of medications that could affect exercise ability, blood biomarkers, or muscle biomarkers, including weight loss medications, statins, oral beta-blockers, performance-enhancing drugs, metformin or other diabetic drug, and oral corticosteroids.
* Use of any sex hormones (estrogen, progesterone, testosterone or other androgens, for the previous 3 months) of any type including oral, creams, vaginal creams or inserts, patches, implants). Participants will be allowed to be on maintenance anti-estrogen therapy - e.g., tamoxifen, aromatase inhibitors
* Consumption of (on average) more than 2 alcoholic drinks per day
* Current use of any tobacco products including smoking, vaping, chew, nicotine patches
* Frequent marijuana use (>1 per month)
* Current participation in another randomized controlled trial

Completed Exclusion Criteria (for participants enrolled prior to Extension portion of study):

* Pregnant in past 3 months
* Lactating
* Premenopausal women: irregular menstrual periods for the previous 6 months; no use of oral contraceptives for the previous 3 months, no use of hormone implants or intrauterine device (IUD) for in the previous year, no use of other sex hormones including testosterone or other androgens for the previous 3 months
* Postmenopausal women: no use of any sex hormones (estrogen, progesterone, testosterone or other androgens, for the previous 3 months) of any type including oral, creams, vaginal creams or inserts, patches, implants
* Current use of any tobacco products including smoking, vaping, chew, nicotine patches
* History of diabetes mellitus, or fasting glucose fingerstick ≥ 126 mg/dL
* Taking any medications to treat high blood sugar such as metformin
* Personal history of invasive or in situ breast cancer
* Personal history of cancer other than breast: exceptions are non-melanoma skin cancer and cervical neoplasia (CIN)
* ≥ 2 alcoholic drinks/day
* Contraindications to exercise
* Abnormalities on screening physical that contraindicate participation
* Contraindications for entry into a research exercise program: recent (within 6 months) myocardial infarction, pulmonary edema, myocarditis, pericarditis, unstable angina, pulmonary embolism, deep vein thrombosis, uncontrolled hypertension (systolic > 200, diastolic > 100), orthostatic hypotension, moderate/severe aortic stenosis, uncontrolled arrhythmia, uncontrolled congestive heart failure, left bundle branch block, history of cardiac arrest or stroke
* Frequent marijuana use (> 1 per month)
* Alcohol or drug abuse, significant mental illness (as assessed by study staff impression)
* History of clotting disorders (muscle-biopsy sub study)
* Unable or unwilling to stop aspirin or nonsteroidal antiinflammatory drugs (NSAIDs) for 48 hours before and after the procedure (muscle-biopsy sub study)
* Allergy to anesthetics or local anesthetics (muscle-biopsy sub study)
* Long term use of warfarin or similar medications (muscle-biopsy sub study)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Mean change in homeostatic model assessment of insulin resistance (HOMA-IR) | Baseline up to 45 minutes
  Will compare the average changes in HOMA-IR from baseline to 45 minutes between the exercisers and controls.
Mean change in HOMA-IR | Baseline up to 105 minutes
  Will compare the average changes in HOMA-IR from baseline to 105 minutes between the exercisers and controls.
Change in insulin level | Baseline up to 45 minutes
  Will compare changes in insulin level from baseline to 45 minutes between the exercisers and controls.
Change in insulin level | Baseline up to 105 minutes
  Will compare changes in insulin level from baseline to 105 minutes between the exercisers and controls.
Change in glucose level | Baseline up to 45 minutes
  Will compare changes in glucose level from baseline to 45 minutes between the exercisers and controls.
Change in glucose level | Baseline up to 105 minutes
  Will compare changes in glucose level from baseline to 105 minutes between the exercisers and controls.
Change in Vascular Endothelial Growth Factor (VEGF) level | Baseline up to 45 minutes
  Will compare changes in VEGF level from baseline to 45 minutes between the exercisers and controls.
Change in VEGF level | Baseline up to 105 minutes
  Will compare changes in VEGF level from baseline to 105 minutes between the exercisers and controls.
Change in Irisin level | Baseline up to 45 minutes
  Will compare changes in Irisin level from baseline to 45 minutes between the exercisers and controls.
Change in Irisin level | Baseline up to 105 minutes
  Will compare changes in Irisin level from baseline to 105 minutes between the exercisers and controls.
Change in Plasminogen activator inhibitor type-1 (PAI-1) level | Baseline up to 45 minutes
  Will compare changes in PAI-1 level from baseline to 45 minutes between the exercisers and controls.
Change in PAI-1 level | Baseline up to 105 minutes
  Will compare changes in PAI-1 level from baseline to 105 minutes between the exercisers and controls.

SECONDARY OUTCOMES:
Effects of exercise on HOMA-IR in normal-weight participants | At 45 minutes
  Will use the generalized estimating equations (GEE) model including the potential effect modification of weight category (normal weight versus [vs] overweight/obese) to compare the 45-minute exercise session on HOMA-IR in normal-weight versus overweight/obese women.
Effects of exercise on HOMA-IR in overweight/obese participants | At 45 minutes
  Will use the GEE model including the potential effect modification of weight category (normal weight versus [vs.] overweight/obese) to compare the 45-minute exercise session on HOMA-IR in normal-weight versus overweight/obese women.
Change in C-reactive protein (CRP) | Baseline up to 105 minutes
  Will compare changes in CRP level from baseline to 105 minutes between the exercisers and controls.
Change in Interleukin (IL)-6 | Baseline up to 105 minutes
  Will compare changes in IL-6 level from baseline to 105 minutes between the exercisers and controls.
Change in Monocyte chemotactic protein (MCP)-1 | Baseline up to 105 minutes
  Will compare changes in MCP-1 level from baseline to 105 minutes between the exercisers and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Anne McTiernan, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duggan C, de Dieu Tapsoba J, Warner J, Dash A, Wang CY, McTiernan A. Effects of acute exercise on inflammatory and metabolic biomarkers in women: a randomized controlled trial. NPJ Breast Cancer. 2025 Nov 7;11(1):122. doi: 10.1038/s41523-025-00834-8. PMID 41203676